CLINICAL TRIAL: NCT06442657
Title: Comparison of Two Care Strategies (5-layer Hydrocellular Dressings Versus Thick Hydrocolloid Dressings) in Preventing the Development of Pressure Sore Lesions Induced by Prone Positioning in Intensive Care Patients. Multicenter Randomized Controlled Trial
Brief Title: Pressure Sore Prevention Strategy for the Prone Position
Acronym: DERM-H-PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A00932-43
Record Dates: First submitted 2024-05-22; First posted 2024-06-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-05

CONDITIONS: Pressure Ulcers Prevention in Prone Positioning in Intensive Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocellular (Experimental): Application of hydrocellular dressings prior to prone positioning and standard pressure sore prevention strategy. Dressings can remain in place for up to 7 days.
  Interventions: Other: Hydrocellular dressing
- Hydrocolloid (Active Comparator): Application of hydrocolloids dressings prior to prone positioning and standard pressure sore prevention strategy. Dressings are removed after each prone position.
  Interventions: Other: Hydrocolloids dressing

INTERVENTIONS:
Other: Hydrocellular dressing — Application of hydrocellular dressings to at-risk areas prior to prone positioning. Assessment of pressure sores and their stage after prone positioning.
  Arms: Hydrocellular
Other: Hydrocolloids dressing — Application of hydrocolloids dressings to at-risk areas prior to prone positioning.
  Arms: Hydrocolloid

SUMMARY:
The aim of this clinical trial is to determine whether 5-layer hydrocellular dressings are effective in preventing the development of pressure sores during prone positioning in the intensive care unit. The main questions it aims to answer are:

- are hydrocellular dressings the best strategy for preventing pressure sores? is this strategy simpler and less costly? The researchers will compare hydrocellular dressings with hydrocolloid dressings to find out whether they are more effective in preventing the development of pressure sores in the prone position.

Participants will be given either hydrocellular or hydrocolloid dressings, and caregivers will assess whether or not pressure sores develop after prone positioning.

DETAILED DESCRIPTION:
Hydrocellular dressings will be compared with hydrocolloid dressings to determine their effectiveness in preventing pressure ulcers during ventral decubitus in intensive care. The dressings will cover the skin in at-risk areas, and caregivers will assess whether or not pressure sores develop in these areas after prone positioning. The stage of these pressure sores will also be assessed.

The time spent on each strategy and the cost per strategy will also be evaluated. Dressings will be applied for the entire period during which participants are placed in the prone position. If they develop pressure sores during this period, they will be followed up until their discharge from intensive care to study the evolution of these pressure sores.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Moderate to severe acute respiratory distress syndrom (Arterial oxygen pressure /Inspired Fraction of oxygen ratio < 200) requiring at least one VD session.
* Affiliated to the French social security system
* Sedated patient on mechanical ventilation

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patient under guardianship or trusteeship
* Minor patients

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Compare the time to onset of one or more pressure ulcers during Ventral Decubitus(VD) sessions in the ICU with the type of preventive dressing selected (thick hydrocolloid or 5-layer hydrocellular) | 30 minutes after being put back on its back
  Time to occurrence of a grade 2 or higher pressure ulcer in the intensive care unit in VD, according to the National Pressure Ulcer Advisory Panel (NPUAP) classification

SECONDARY OUTCOMES:
Compare the location of pressure sores between the two groups | 30 minutes after putting the participant back on his back
  Number of pressure sores (stages 1 to 4) on predetermined risk areas protected by both types of dressing (periorbital, malar, mandible/chin, thorax, shoulders, iliac crests, knees, other).
Compare the severity of pressure sores between the two groups | 30 minutes after putting the participant back on his back
  Severity of pressure sore according to NPUAP classification (stages 1 to 4)
Compare the evolution of pressure sores between the two groups up to discharge from the intensive care unit. | 30 minutes after the participant has been put back on his back after each prone session, then at D7, D14 and D28 or at discharge from intensive care if the participant has had a pressure sore
  Evolution of the pressure sore according to NPUAP classification. During the VD period, assessment is carried out daily after repositioning in Dorsal Decubitus (DD). After the end of the DV, any dressings applied to treat a pressure sore will no longer be the randomized dressings, but the most suitable dressings according to the predefined management protocol . Classification of the pressure sore will be carried out at D7, D14, D28 or on the day of discharge from the intensive care unit
Compare the care required to apply, monitor and remove the two types of dressing | Three years
  Time spent on each of the two care strategies in minutes
Compare the cost of medical devices, by dressing strategy, until VD sessions are discontinued | Three years
  Overall cost of each care strategy. An assessment of the direct cost of dressings will be made on the basis of the number recorded for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Agathe Hamelin, Principal Investigator — CHU CAEN
Locations (1):
- CHU, Caen, France

IPD SHARING:
Plan to Share IPD: No